CLINICAL TRIAL: NCT04499417
Title: Psychological and Physical Effects of an 8-Week Electromyostimulation-Whole-Body-Workout
Brief Title: Psychological and Physical Effects of an 8-Week Electromyostimulation-Workout
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: miha bodytec GmbH (Unknown)
Responsible Party: Principal Investigator, Antonia Bendau, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA4/058/19 (longterm trial)
Record Dates: First submitted 2020-07-26; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Physical Activity; Exercise; Mental Health; Health Behaviour; Electromyostimulation; EMS; Strength Training
MeSH Terms: conditions — Motor Activity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study has a randomised placebo-controlled parallel design (two arms: experimental-condition, sham-condition).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and Outcomes Assessors are not aware of the study hypothesis / the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-Condition (Experimental): 8 weeks x weekly 20 minutes whole-body-workouts with simultaneous muscle stimulation (EMS).
  Participants carry out easy whole-body-exercises while wearing a EMS-vest-belt-system with interwoven electrodes. During the workout the muscles are simultaneously stimulated by those external electrodes with medium level (5) of stimulation intensity.
  Interventions: Device: Electromyostimulation Whole-Body-Workout
- Sham-Condition (Sham Comparator): 8 weeks x weekly 20 minutes whole-body-workouts without simultaneous muscle stimulation (EMS).
  Participants carry out easy whole-body-exercises while wearing a EMS-vest-belt-system with interwoven electrodes. During the workout the muscles are not actually stimulated by EMS.
  Interventions: Device: Electromyostimulation Sham Whole-Body-Workout

INTERVENTIONS:
Device: Electromyostimulation Whole-Body-Workout — Electromyostimulation - intensity 5 (muscle stimulation)
  Other Names: EMS
  Arms: Experimental-Condition
Device: Electromyostimulation Sham Whole-Body-Workout — Electromyostimulation - intensity 0 (no muscle stimulation)
  Other Names: EMS-Sham
  Arms: Sham-Condition

SUMMARY:
The study investigates the midterm, longterm and acute psychological and physical effects of an 8-week whole-body-workout using Electromyostimulation (EMS) in healthy individuals.

DETAILED DESCRIPTION:
EMS-whole-body-workouts are less time-consuming and effort-intensive but generate physical effects which are comparable to conventional strength training. Therefore EMS could lower the barrier to physical activity. The present study focusses on psychological and physical effects of an 8-week EMS workout. Physical activity is notably important for mental and physical health, but is on average far too rarely implemented. Therefore EMS-whole-body-workouts could provide an opportunity to generate positive psychological and physical effects through a less (subjective) cost-intense strength training.

ELIGIBILITY:
Inclusion Criteria:

* Subject familiarized with experimental procedure and had given written informed consent
* Able to understand German
* Reachability of participant for the eight training sessions

Exclusion Criteria:

* Contraindications for physical exercise or EMS-use
* Current EMS-use or intense regular exercise (> 60 min / week)
* Pregnancy
* Current presence of any mental disease
* Acute suicidality
* Substance dependencies with actual consumption (except nicotine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-07-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Acute change of subjective well-being. | From directly before each of the eight training sessions do directly after each of the sessions (EMS-Training/Sham) during the 8 weeks of training.
  • Subjective well-being is measured using a visual analogue scale (0-100%, higher value = better outcome).
Acute change of subjective relaxation. | From directly before each of the eight training sessions do directly after each of the sessions (EMS-Training/Sham) during the 8 weeks of training.
  • Subjective relaxation is measured using a visual analogue scale (0-100%, higher value = better outcome).
Change of acute symptoms of anxiety and depression. | From directly before each of the eight training sessions do directly after each of the sessions (EMS-Training/Sham) during the 8 weeks of training.
  • The State-Scale of the State-Trait-Anxiety-Depression-Inventar (STADI-State; Renner, Hock, Bergner-Köther & Laux, 2018) is used to assess acute symptoms of depression and anxiety. The raw score ranges from 10 to 40, higher values indicate a worse outcome.

SECONDARY OUTCOMES:
Mid-/longterm changes in depressive symptoms. | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • Patient Health Questionnaire (PHQ-9; Kroenke & Spitzer, 2002). Sum scores ranging from 0 to 27, higher values indicate a worse outcome.
Mid-/longterm changes in anxiety symptoms. | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • Generalized Anxiety Disorder Scale (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006). Sum scores ranging from 0 to 21, higher values indicate a worse outcome.
Mid-/longterm changes in affect-related psychological variables. | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • The Trait-Scale of the State-Trait-Anxiety-Depression-Inventar (STADI-Trait; Renner, Hock, Bergner-Köther & Laux, 2018) is used to assess symptoms of depression and anxiety. The raw score ranges from 10 to 40, higher values indicate a worse outcome.
Mid-/longterm changes in positive and negative affect. | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • Positive and Negative Affect Schedule (PANAS; Watson, Clark & Tellegen, 1988). Positive subscale: Scores ranging from 10 to 50, higher scores represent a better outcome. Negative subscale: Scores ranging from 10 to 50, higher scores represent a worse outcome.
Change in general self-efficacy | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • General self-efficacy is measured using the General-Self-Efficacy Scale (GSE) by Jerusalem & Schwarzer (1981). The GSE has 10 likert scaled items with values ranging from 1 to 4, higher scores mean a better outcome.
Change in attitudes regarding physical activity (intentions for physical activity, self-efficacy regarding physical activity) | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • Intention (4 items) and self-efficacy (2 items) are measured using six likert scaled items by Petzold et al. (2017). Values ranging from 1 to 4, higher scores mean a better outcome.
Change in physical parameters: heart rate variability. | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • Heart rate variability is measured with a polar chest strap during 5 minutes of relaxation.
Change in physical parameters: hand force. | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • Hand force is measured with a hand-dynamometer left and right hand.
Change in physical parameters: leg strength. | Baseline (before any training) + Intermediate (4 weeks) + Post (8 weeks) + Follow-Up (12 weeks).
  • Leg strength is assessed using the 30-second chair-stand-test.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof.Dr., Study Director — Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy; Antonia Bendau, M.Sc.Psych., Principal Investigator — Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy
Locations (1):
- Charité-Universitätsmedizin Berlin - Department of Psychiatry and Psychotherapy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No